CLINICAL TRIAL: NCT03175653
Title: Assessing the Impact of the Number of Opiates Prescribed on Post Cesarean Pain Control: A Randomized Controlled Trial
Brief Title: Impact of the Number of Opiates Prescribed on Post Cesarean Pain Control
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility - could not operationalize prior to PI leaving the institution.
Sponsor: Mount Carmel Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 170214-2
Record Dates: First submitted 2017-05-04; First posted 2017-06-05 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2020-09

CONDITIONS: Post-operative Pain Control
MeSH Terms: interventions — Oxycodone

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Masking Description: Participants and investigators will be aware of the arm to which they have been assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A - Oxycodone Pill A (Experimental): Participants in this study arm will receive a prescription for a lower number oxycodone (oxycodone A) pills for post-cesarean pain control.
  Interventions: Other: Oxycodone Pill A
- Arm B - Oxycodone Pill B (Active Comparator): Participants in this study arm will receive a prescription for a higher number of oxycodone (oxycodone B) pills for post-cesarean pain control.
  Interventions: Other: Oxycodone Pill B

INTERVENTIONS:
Other: Oxycodone Pill A — Prescription for oxycodone pills for post-Cesarean delivery pain control after hospital discharge. Oxycodone is an opioid.
  Other Names: Oxycodone pill - lower number
  Arms: Arm A - Oxycodone Pill A
Other: Oxycodone Pill B — Prescription for oxycodone pills for post-Cesarean delivery pain control after hospital discharge. Oxycodone is an opioid.
  Other Names: Oxycodone pill - higher number
  Arms: Arm B - Oxycodone Pill B

SUMMARY:
The purpose of this randomized trial is to examine whether the number of opioid pills prescribed for pain control after Cesarean section has an effect on patient reported pain levels and satisfaction with pain control during recovery. Both groups receive what is considered an adequate number of pills for pain control after an uncomplicated Cesarean delivery. Secondarily, the investigators wish to gather reliable information about the duration of use of opioids for pain control after uncomplicated Cesarean section, and what happens to unused medication.

After an uncomplicated Cesarean section, patients will be approached and asked to participate in the study. If the patient agrees, she will be randomly assigned to one of the two study groups and receive a prescription for opioid medication at the time of hospital discharge. At her standard care follow-up visit 10-14 days later, the participant will complete a survey asking questions about her pain levels during recovery, her use of study-related and non-study-related pain medication, and satisfaction with pain control. At that point the patient's participation in the study will end.

DETAILED DESCRIPTION:
Study Design and Methods:

The investigators will conduct a randomized controlled trial evaluating the difference in postpartum pain control in women receiving two different amounts of oxycodone after cesarean delivery.

Primary outcomes

• The primary outcome is the percent of patients who refill their narcotic prescription after cesarean delivery.

Secondary outcomes

1. Duration of use of narcotic after cesarean delivery, as assessed by the Post Cesarean Pain Control Survey (see attachment).
2. Amount of narcotic unused after cesarean delivery, measured in number of remaining pills, as assessed by the Post Cesarean Pain Control Survey.
3. Disposition of unused drug, as assessed by the Post Cesarean Pain Control Survey.
4. Patient satisfaction with pain control after cesarean delivery, as assessed by the Post Cesarean Pain Control Survey.

Patients will be identified by one of the investigators or designated research staff as either scheduled to undergo repeat cesarean delivery or status post cesarean from review of postpartum delivery lists. If they meet inclusion and exclusion criteria, they will be approached for enrollment in the study. If they consent they will be randomized on the day of discharge to group A or group B via sequentially numbered, sealed, opaque envelope. All patients will be provided standard education regarding pain control in the form of a fact sheet regarding trajectories of pain resolution, normative opioid consumption post cesarean, as well as risks, benefits and alternatives to opiates. If unable to purchase over the counter medications, prescriptions for ibuprofen and acetaminophen will be provided, as well as phone numbers for contact should any concerns arise between the time of discharge and post operative assessment. The patient will be scheduled for a postoperative wound check 10-14 days postpartum.

Postoperative wound evaluation will be performed in the research site's OB clinic setting at which time the survey will be completed by the patient regarding satisfaction with pain control, length of opiate treatment, number of opiates left in prescription and need for refills.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-45 years
* English, Somali or Spanish Speaking
* Status post uncomplicated cesarean delivery performed at term (37w 0d to 42w 0d at time of delivery)
* Discharged at day 3 or 4 after cesarean section
* Willingness to participate in a survey 10-14 days post cesarean

Exclusion Criteria:

* History of or current narcotic abuse
* History of chronic pain
* History or current opiate addiction
* Complicated cesarean delivery including cesarean hysterectomy, EBL >1500 cc, bowel or bladder injury, postpartum infectious morbidity, postpartum wound break down
* Neonatal outcome requiring NICU admission for more than 48 hours

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females who self-identify, are able to get pregnant and who undergo Cesarean section.
Enrollment: 0 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the percent of patients who refill their narcotic prescription after cesarean delivery. . | 7-14 days after surgery
  This outcome will be assessed by survey and confirmed with Ohio Automatic Rx Reporting System (OARRS) review performed on the same day as survey completion

SECONDARY OUTCOMES:
Duration of use of narcotic after cesarean | 7-14 days after surgery
  As assessed by the Post Cesarean Pain Control Survey
Amount of narcotic unused after cesarean delivery. | 7-14 days after surgery
  Measured in number of remaining pills, as assessed by the Post Cesarean Pain Control Survey
Disposition of unused drug | 7-14 days after surgery
  As assessed by the Post Cesarean Pain Control Survey.
Patient satisfaction with pain control after cesarean delivery | 7-14 days after surgery
  As assessed by the Post Cesarean Pain Control Survey.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Prasad, DO, Principal Investigator — Mount Carmel Health System
Locations (1):
- Mt Carmel Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reddy UM. Screening, Prevention, and Treatment of Opioid Use Disorder During Pregnancy: Expectant Mothers Are Depending on You! Obstet Gynecol. 2016 Jul;128(1):1-3. doi: 10.1097/AOG.0000000000001505. No abstract available. PMID 27275810
- [Background] Krans EE, Patrick SW. Opioid Use Disorder in Pregnancy: Health Policy and Practice in the Midst of an Epidemic. Obstet Gynecol. 2016 Jul;128(1):4-10. doi: 10.1097/AOG.0000000000001446. PMID 27275812
- [Background] Pfuntner A, Wier LM, Stocks C. Most Frequent Procedures Performed in U.S. Hospitals, 2011. 2013 Oct. In: Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Statistical Brief #165. Available from http://www.ncbi.nlm.nih.gov/books/NBK174682/ PMID 24354027
- [Background] 1. Osmundson, S, Grasch JL, Schornack LA, et al. Opioid Use after cesarean delivery following hospital discharge. American Journal of Obstetrics and Gynecology, 2017. 216:1(Supplement 1): Abstract 704, S411-S412.